CLINICAL TRIAL: NCT03732092
Title: The Effects of Olfactory Stimulation on Diagnosis and Prognosis of Patients With Disorders of Consciousness
Brief Title: The Effects of Olfactory Stimulation on Diagnosis and Prognosis of DOC Patients
Status: Completed | Type: Observational
Sponsor: Jing Wang (Other)
Responsible Party: Sponsor-Investigator, Jing Wang, Principal Investigator, Hangzhou Normal University
Organization: Hangzhou Normal University (Other)
Other Study IDs: 2018A04355
Record Dates: First submitted 2018-11-04; First posted 2018-11-06 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Minimally Conscious State; Vegetative State
Keywords: disorders of consciousness; prognosis prediction; minimally conscious state; vegetative state; olfactory stimulation
MeSH Terms: conditions — Persistent Vegetative State; Consciousness Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with disorders of consciousness: Patients with disorders of consciousness from several brain injury, assessed by Coma Recovery Scale-Revised (CRS-R), have been clinically classified into coma, unresponsive wakefulness syndrome and minimally conscious state.
  Interventions: Diagnostic Test: Coma Recovery Scale-Revised

INTERVENTIONS:
Diagnostic Test: Coma Recovery Scale-Revised — Patients with disorders of consciousness were assessed by Coma Recovery Scale-Revised (CRS-R). In addition, we selected three stimuli: 1) 1-octene-3-ol, 2) pyridine, 3) water. We presented these three stimuli in front of the patients nose for 3 seconds.

SUMMARY:
Analyze the behavioral response of patients with disorders of consciousness through olfactory stimulation, compare the response of olfactory stimulation in patients with different consciousness, and analyze the impact of olfactory stimulation on diagnosis; After the first, third, and sixth months of initial enrollment, the recovery of prognosis was tracked by the Coma Recovery Scale-Revision (CRS-R).

DETAILED DESCRIPTION:
Previous studies suggested that olfactory stimulus have some effect on some patients with disorders of consciousness. Then, the aim of the present study is to know the prognostic value of olfactory stimulation and the diagnosis for DOC patients. DOC patients were recruited (standard diagnosis procedure is 5 times CRS-R testing within 10 days). The different stimuli were as follows: 1) 1-octene-3-ol, odor. 2) pyridine, odor. 3) water. We presented these stimuli randomly, and we recorded the patient's CRS-R scale behavioral response and response to olfactory stimulation. Analyze the behavioral response of patients with disorders of consciousness through olfactory stimulation, compare the response of olfactory stimulation in patients with different consciousness, and analyze the impact of olfactory stimulation on diagnosis; After the first, third, and sixth months of initial enrollment, the recovery of prognosis was tracked by the Coma Recovery Scale-Revision (CRS-R).

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old;
* non-acute phase;
* after coma;
* no nerve stimulation drugs within 48 hours before the implementation of the study;
* no neuromuscular blockers within 24 hours before implementation

Exclusion Criteria:

* history of forehead injury;
* nasal fractures;
* tracheotomy;
* developmental mental or neurological diseases leading to recorded dysfunction;
* severe fractures of the extremities.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with disorders of consciousness
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Coma Recovery Scale-Revised （CRS-R） | six months later
  The CRS-R consists of 23 items grouped in six subscales addressing auditory, visual, motor, oromotor, communication and arousal functions. The higher items represent conscious related behaviour while the lower items for each sub-scale represent reflexive activity. Basis for scoring was the presence or absence of the specific behaviour in response to standard stimuli. Patients were followed up for 1, 3, and 6 months to track the prognosis of patients by CRS-R.

CONTACTS AND LOCATIONS:
Overall Officials: Patients with disorders of consciousness were assessed by Coma Di, Pro, Study Chair — International Vegetative State and Consciousness Science Institute, Hangzhou Normal University
Locations (1):
- International Vegetative State and Consciousness Science Institute, Hangzhou Normal University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Chiaravalloti A, Pagani M, Micarelli A, Di Pietro B, Genovesi G, Alessandrini M, Schillaci O. Cortical activity during olfactory stimulation in multiple chemical sensitivity: a (18)F-FDG PET/CT study. Eur J Nucl Med Mol Imaging. 2015 Apr;42(5):733-40. doi: 10.1007/s00259-014-2969-2. Epub 2015 Feb 18. PMID 25690545
- [Derived] Wang J, Zhang S, Liu W, Zhang Y, Hu Z, Sun Z, Di H. Olfactory Stimulation and the Diagnosis of Patients With Disorders of Consciousness: A Double-Blind, Randomized Clinical Trial. Front Neurosci. 2022 Feb 17;16:712891. doi: 10.3389/fnins.2022.712891. eCollection 2022. PMID 35250440